CLINICAL TRIAL: NCT01697059
Title: Initial Antibiotics and Delayed Appendectomy for Acute Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Francois Luks, Francois I. Luks, MD, PhD, Rhode Island Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIH408212
Record Dates: First submitted 2012-09-24; First posted 2012-10-02 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Acute Appendicitis
Keywords: appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Piperacillin; Amoxicillin; Piperacillin, Tazobactam Drug Combination; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Piperacillin + Amoxicillin (Experimental): Piperacillin/Tazobactam (Zosyn®) 100 mg/kg, up to adult dose of 3 g, i.v. q 6 hours x 2 doses, followed by Ampicillin/Clavulanate (Augmentin®) 50 mg/kg/d p.o. in 3 divided doses for 1 week.
  Interventions: Drug: Piperacillin + Amoxicillin

INTERVENTIONS:
Drug: Piperacillin + Amoxicillin
  Other Names: Zosyn®; Augmentin®

SUMMARY:
Several recent studies have examined the feasibility and benefits of nonoperative treatment of perforated appendicitis in children. One such study showed a trend toward longer operative times for patients randomized to immediate appendectomy, but no overall advantage. In another larger study, the costs of delayed appendectomy for perforated appendicitis were higher - in part related to readmissions in the interval (6-8 weeks). Nevertheless, these and other studies have demonstrated the safety of delaying appendectomy for perforated appendicitis.

Emergency appendectomy is a well-established approach, and postoperative recovery in children is fast. Nevertheless, from the onset of symptoms through the hospital stay and the postoperative recovery, appendicitis causes a disruption of a family's normal routine (absence from school and work) of up to 1-2 weeks. Because this is an unplanned operation, patients have to wait until an operating room becomes available, or elective operations have to be placed on hold to accommodate the emergency operation. Each year, more than 250 children undergo an appendectomy at HCH. This represents 250 episodes of emergency surgery, or about one emergency add-on operation per working day. If an initial trial of antibiotics is safe for the treatment of appendicitis, converting an emergency operation into an elective, scheduled outpatient procedure may reduce stress and disruption of routine for patients and their families - and may allow better operating room planning for health care professionals and hospitals.

The investigators hypothesize that initial antibiotic treatment of acute (non-perforated) appendicitis, followed by scheduled outpatient appendectomy, reduces the overall cost of treating the disease and results in greater patient and family satisfaction.

This pilot study aims to establish the safety and feasibility of treating acute appendicitis with intravenous antibiotics, followed by outpatient oral antibiotics. Patients and their families will be offered the possibility of initial nonoperative treatment and subsequent outpatient elective appendectomy in a nonrandomized, single arm study.

ELIGIBILITY:
Inclusion Criteria:

* Maximum 48-hour-history of abdominal pain
* Diagnosis of acute appendicitis based on clinical, laboratory and/or radiologic criteria

Exclusion Criteria:

* Duration of symptoms > 48 hours
* Presence of an appendiceal abscess on imaging
* Clinical or laboratory suspicion of advanced appendicitis, peritonitis or perforation
* Significant comorbidities
* Inability or unwillingness to complete a 1-week course of oral antibiotics
* Allergy to penicillin

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of treatment failures | Worsening of symptoms at 8 hours or failure of improvement at 18 hours of treatment
  If after a period of at least 8 hours (and 2 doses of intravenous antibiotics), the patient's symptoms worsen, or fail to subside within 18 hours, the patient will undergo an emergent/urgent appendectomy, and treatment will proceed as per standard-of-care (1 intraoperative dose of antibiotics, with or without postoperative antibiotics, progressive postoperative diet and discharge home once tolerating a regular diet). The patient will then be considered having failed nonoperative treatment.

SECONDARY OUTCOMES:
Cost-saving of initial nonoperative treatment for early appendicitis | 1 year
  Cost of nonoperative treatment will be calculated as follows: Hospitalization charges (# hospital days - observation) + costs of antibiotics (actual number of doses/days) + outpatient surgery hospital fee (operating room and PACU time) + additional costs associated with unanticipated events (e.g., Emergency room visits after initial discharge).
  Control costs (contemporary data) will consider the following: Hospitalization charges (# hospital days) + intravenous antibiotics (price/dose x number of doses).

OTHER OUTCOMES:
Utility of initial nonoperative treatment of early appendicitis | 1 year
  Questionnaires given to parents and patients regarding their experience of initial nonoperative treatment and interval appendectomy will be analyzed, and compared with controls and with standard levels in the literature.
  The Pediatric Quality of Life Scale-Version 4.0 (PedsQL) is a reliable and valid 23-item questionnaire that measures child health-related quality of life (QOL) in the preceding month. Items can be recoded from 100 to 0 on 25-point intervals and averaged to produce a total score (α=0.90). The total score is derived from items that assess the child's physical (e.g., problems with low energy or difficulty lifting something heavy), emotional (e.g., feeling afraid, angry, or scared), social (e.g., problems with getting teased or other children not wanting to be friends), and school functioning (e.g., problems paying attention in class or missing school). Higher scores indicate better QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Francois I. Luks, MD, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Hasbro Children's Hospital (Rhode Island Hospital), Providence, Rhode Island, United States

REFERENCES:
- [Background] Narsule CK, Kahle EJ, Kim DS, Anderson AC, Luks FI. Effect of delay in presentation on rate of perforation in children with appendicitis. Am J Emerg Med. 2011 Oct;29(8):890-3. doi: 10.1016/j.ajem.2010.04.005. Epub 2010 Jul 13. PMID 20627213
- [Background] Powers RJ, Andrassy RJ, Brennan LP, Weitzman JJ. Alternate approach to the management of acute perforating appendicitis in children. Surg Gynecol Obstet. 1981 Apr;152(4):473-5. PMID 7209777
- [Background] St Peter SD, Aguayo P, Fraser JD, Keckler SJ, Sharp SW, Leys CM, Murphy JP, Snyder CL, Sharp RJ, Andrews WS, Holcomb GW 3rd, Ostlie DJ. Initial laparoscopic appendectomy versus initial nonoperative management and interval appendectomy for perforated appendicitis with abscess: a prospective, randomized trial. J Pediatr Surg. 2010 Jan;45(1):236-40. doi: 10.1016/j.jpedsurg.2009.10.039. PMID 20105610
- [Background] Styrud J, Eriksson S, Nilsson I, Ahlberg G, Haapaniemi S, Neovius G, Rex L, Badume I, Granstrom L. Appendectomy versus antibiotic treatment in acute appendicitis. a prospective multicenter randomized controlled trial. World J Surg. 2006 Jun;30(6):1033-7. doi: 10.1007/s00268-005-0304-6. PMID 16736333
- [Background] Yardeni D, Hirschl RB, Drongowski RA, Teitelbaum DH, Geiger JD, Coran AG. Delayed versus immediate surgery in acute appendicitis: do we need to operate during the night? J Pediatr Surg. 2004 Mar;39(3):464-9; discussion 464-9. doi: 10.1016/j.jpedsurg.2003.11.020. PMID 15017571